CLINICAL TRIAL: NCT07293767
Title: The Effect of Silymarin Versus Hesperidin/Diosmin Combination on Patients With Fibromyalgia
Brief Title: Silymarin vs Hesperidin/Diosmin in Fibromyalgia
Acronym: SHD-FM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, minna sayed, pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FM
Record Dates: First submitted 2025-11-25; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Fibromyalgia (FM)
Keywords: fibromyalgia; silymarin; hesperidin; diosmin
MeSH Terms: conditions — Fibromyalgia | interventions — Silymarin; Diosmin; Hesperidin; Control Groups

STUDY DESIGN:
Intervention Model Description: Group I: 30 patients will receive their standard treatment of fibromyalgia for four months. Group II: 30 patients will receive 500 mg of diosmin/ hesperidine combination under the trade name of daflon with their standard treatment of fibromyalgia for four months. Group III: 30 patients will receive 140 mg of silymarin three times daily under the trade name of Legalon with their standard treatment for four months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Silymarin group (Experimental): this group of patients will receive silymarin (LEGALON) 140 mg three times daily with the standard treatment
  Interventions: Drug: Silymarin (LEGALON)
- Diosmin/hisperedin group (Experimental): this group will receive hesperidin/diosmin (daflon) 500 once daily for 12 weeks with the standard treatment
  Interventions: Drug: Diosmin / Hesperidin (Daflon)
- Standard care group (Active Comparator): participants will receive standard treatment only
  Interventions: Other: no intervention (control group)

INTERVENTIONS:
Drug: Silymarin (LEGALON) — oral silymarin (legalon) 140 mg will be taken 3 times daily for 12 weeks with the standard treatment
  Arms: Silymarin group
Drug: Diosmin / Hesperidin (Daflon) — Diosmin / Hesperidin (Daflon) 500 mg will be taken once daily for 12 weeks with the standard treatment
  Arms: Diosmin/hisperedin group
Other: no intervention (control group) — this group will receive no intervention (only the standard treatment)
  Arms: Standard care group

SUMMARY:
Fibromyalgia is a chronic disease, characterized by chronic widespread pain, physical exhaustion, sleep problems, and unexplained pain in both joints and muscles. Fibromyalgia's causes still unknown, but there are various risk factors that can cause fibromyalgia such as genetic causes, physical shock, and infections. Fibromyalgia typically presents in young or middle aged females, it occurs in females more than males, and it is characterized with widespread pain throughout the whole body in both sides such as arms, shoulders, head, and abdominal areas. The etiology of fibromyalgia still unclear, but there are several factors such as alterations in the sleep pattern, changes in the neuroendocrine transmitters such as cortisol, growth hormones and serotonin, dysfunction of central and autonomic nervous systems, psychiatric aspects and external stressors . The pain seems to result from neurochemical imbalances in the central nervous system that lead to a "central amplification" of pain perception characterized by allodynia (a heightened sensitivity to stimuli that are not normally painful) and hyperalgesia (an increased response to painful stimuli). this interventional study aims to study effect of silymarin and hesperidin/diosmin combination on fibromyalgia patients and compare their effect with control patients on the following

1. Management of pain.
2. Inflammatory biomarkers.
3. Quality of life.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic disease characterized by chronic widespread pain, physical exhaustion, sleep problems, and unexplained pain in joints and muscles. Although the exact causes remain unknown, several risk factors have been implicated, including genetic predisposition, physical or emotional stress, and infections. Fibromyalgia occurs predominantly in females and is associated with widespread pain in multiple body regions such as the arms, shoulders, head, and abdomen. The etiology involves alterations in sleep patterns, changes in neuroendocrine transmitters such as cortisol, growth hormone, and serotonin, along with dysfunction of the central and autonomic nervous systems. Pain is believed to result from neurochemical imbalances that lead to central amplification of pain perception, characterized by allodynia and hyperalgesia.

Diagnosis of fibromyalgia is challenging, as no specific laboratory tests or imaging confirm the condition. The 1990 ACR criteria relied on tender points and widespread pain for at least three months. More recently, the ACR proposed new diagnostic criteria incorporating the Widespread Pain Index (WPI) and Symptom Severity (SS) scale, which evaluate pain in 19 body regions and rate associated symptoms such as fatigue, cognitive difficulties, headache, and dizziness.

Management of fibromyalgia includes several approaches. FDA-approved medications include pregabalin, duloxetine, and milnacipran, although these may be costly and associated with side effects. Anticonvulsants, amitriptyline, and fluoxetine may also be used to improve pain and sleep. Non-pharmacological therapies include biofeedback, cognitive behavioral therapy, physiotherapy, exercise, and electromyogram-guided interventions. Alternative therapies such as acupuncture, chiropractic care, deep tissue massage, neuromuscular massage, meditation, and certain herbal supplements (e.g., echinacea purpurea, black cohosh, lavender, Silybum marianum) have shown varying degrees of benefit.

Inflammatory mediators, particularly IL-6 and IL-8, are commonly elevated in fibromyalgia and correlate with functional impairment, fatigue, and sleep disturbance. Silymarin, extracted from Silybum marianum, possesses hepatoprotective, antioxidant, anti-inflammatory, immunomodulatory, and cardioprotective activities. It has demonstrated reductions in inflammatory cytokines such as TNF-α and IL-6 and showed significant reduction of IL-1α and IL-8 in clinical studies. Diosmin/hesperidin, a flavonoid combination derived from citrus fruits, also exhibits antioxidant and anti-inflammatory activity and has produced antihyperalgesic effects in neuropathic pain models through the reduction of TNF-α, IL-1β, and IL-6.

Based on these findings, the current study hypothesizes that administering silymarin or diosmin/hesperidin in addition to standard fibromyalgia therapy may reduce inflammation and improve pain outcomes in patients with fibromyalgia. The study will compare the effects of silymarin versus diosmin/hesperidin on clinical symptoms, inflammatory biomarkers, and quality of life over a four-month period, as well as evaluate their safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent.
* Participant must meet the American College of Rheumatology 2016 revised classification criteria for Fibromyalgia: Widespread pain index (WPI) ≥ 7 and symptom severity (SS) scale score ≥ 5, or WPI 3 to 6 and SS scale score ≥ 9
* Age >18 years old (males and females)
* Diagnosis of FM confirmed by a rheumatologist.
* Persistent pain syndrome on conventional therapy.
* Not taking Daflon or Legalon for 6 months.

Exclusion Criteria:

* Pain due to other conditions (e.g. diabetic peripheral neuropathic pain or post-herpetic neuralgia) that would confound assessment or self-evaluation of the pain associated with FM.
* Patients with pain due to any widespread inflammatory musculoskeletal disorder (e.g. rheumatoid arthritis, lupus) or widespread rheumatic disease other than FM.
* Allergy to silymarin or diosmin or hesperidin.
* Cognitive deficits that could impair understanding of the study, completion of questionnaires, or adherence to therapy.
* Pregnant or planning pregnancy women and breastfeeding women.
* Major comorbidities like renal impairment, severe liver disease, chronic hepatitis C, history of alcohol or drug addiction.
* Current severe or uncontrolled major depressive disorder or anxiety disorders.
* Patients will be excluded if there is no compliance to the medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-16 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
pain assessment through Fibromyalgia impact questionnaire (FIQ) | 4 months
  Change in Fibromyalgia impact questionnaire (FIQ) score will be assessed by the end of the study, the score ranges from 0 to 100 higher score means worse condition

SECONDARY OUTCOMES:
Erythrocyte sedimentation rate (ESR) | 4 months
  ESR will be measured at baseline and after four months of treatment
C-reactive protein level (CRP) | 4 months
  CRP will be measured at baseline and after four months of treatment
Health-related quality-of-life through Short Form 12 health survey SF-12 | 4 months
  quality of life will be assessed through Short Form 12 health survey SF-12 (Questionnaire of health) at baseline and after 4 months the score ranges from 0 to 100 higher scores indicate better health
pain assessment through visual analogue scale (VAS) | 4 months
  visual analogue scale (VAS) score will be assessed at baseline and after four months of treatment, the score ranges from 0 to 10 cm higher score means worse condition
laboratory evaluation of interleukin- 8 (IL-8) level | 4 months
  serum IL8 concentration will be measured at baseline and after four months of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatients clinic of department of Internal medicine- Rheumatology unit Ain shams hospitals., Cairo, Egypt